CLINICAL TRIAL: NCT00558831
Title: A Split-face, Paired-comparison Pilot Study to Evaluate the Safety and Efficacy of Topical Benzoyl Peroxide 2.5% Cream Alone Versus Benzoyl Peroxide 2.5% Cream Plus Moisturizing Lotion for Mild to Moderate Acne Vulgaris
Brief Title: Study of Benzoyl Peroxide Cream for Mild to Moderate Acne Vulgaris
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Amy Paller, Principle Investigator, Northwestern University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU1884
Record Dates: First submitted 2007-11-13; First posted 2007-11-15 (Estimated); Results first posted 2010-11-22 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-08

CONDITIONS: Acne Vulgaris
Keywords: Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — Benzoyl Peroxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Benzoyl Peroxide (Active Comparator): Benzoyl Peroxide (BP) 2.5%
  Interventions: Drug: Benzoyl Peroxide
- Benzoyl Peroxide plus moisturizing lotion (Active Comparator): Benzyol Peroxide 2.5% plus moisturizing lotion
  Interventions: Drug: Benzoyl Peroxide; Drug: Moisturizing Lotion

INTERVENTIONS:
Drug: Benzoyl Peroxide — Benzoyl Peroxide 2.5%
Drug: Moisturizing Lotion
  Arms: Benzoyl Peroxide plus moisturizing lotion

SUMMARY:
The purpose of this study is to compare the efficacy of a benzoyl peroxide 2.5% cream formulation plus a moisturizing lotion versus benzoyl peroxide 2.5% cream alone for the treatment of acne vulgaris.

DETAILED DESCRIPTION:
The purpose of this study is to compare the safety and efficacy of a benzoyl peroxide 2.5% cream formulation plus a moisturizing lotion versus benzoyl peroxide 2.5% cream alone for mild to moderate acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects who are 18 to 35 years of age.
2. Subjects are in good health and are free of any other facial skin disorders that may interfere with acne study assessments.
3. Subjects have the willingness and ability to understand and provide informed assent/consent to participate in the study and are able to communicate with the investigator. Subjects are willing and able to follow all study directions and to commit to all follow-up visits for the duration of the study. In addition, subjects must be willing to accept the restrictions of the study.
4. A minimum of 2 but no more than 30 inflammatory lesions (papules and pustules), relatively symmetrical in appearance on both sides of the face and a minimum of 2 but not more than 100 non-inflammatory lesions (open comedones and closed comedones) relatively symmetrical in appearance on both sides of the face.
5. Ongoing oral medications (other than those specifically for acne) are acceptable provided subjects are on a stable regimen throughout the study and provided the medications are determined likely to not interfere with study assessments.
6. Subjects will not use medicated cosmetics and/or soaps (including soaps containing antibacterial agents such as benzoyl peroxide, keratolytic agents such as salicylic acid, skin fresheners/astringents or aftershave lotions) for the duration of the study.
7. Subjects who agree not use any other acne treatment (including prescription and non-prescription medications) on the test site for the duration of the study.
8. Subjects who agree not to change facial cosmetic products during the study.
9. Subjects who agree to only use sunscreen/sunblock agents that are labeled as non-comedogenic.

Exclusion Criteria:

1. Subjects or parents of subjects who are unable to understand the protocol or to give informed consent/assent.
2. Subjects with mental illness.
3. Subjects with no inflammatory acne.
4. Subjects with any acne cysts or nodules.
5. Subjects with acne conglobata, acne fulminans, secondary acne (e.g. Chloracne, drug-induced acne), or any acne requiring systemic treatment.
6. Subjects with excessive facial hair that may interfere with study assessments.
7. Subjects with other facial skin disorders that may interfere with study assessments.
8. Subjects with a history of skin cancer or actinic keratosis.
9. Subjects who have used tanning devices within one week prior to baseline study visit.
10. Subjects who have applied any topical products (e.g. emollients, sunscreens) or any cosmetics to the face at least one hour prior to study assessments.
11. Use of hormonal oral contraceptives for acne control or for less than 6 months prior to study baseline.
12. Subjects with known allergies, a history of, or sensitive to salicylic acid, benzoyl peroxide or any of the test article components.
13. Subjects using topical or systemic medication within 14 days before the study entry, which could interfere with study assessments. This includes but is not limited to the following: anti-inflammatory drugs (e.g. topical and systemic corticosteroids and systemic antihistamines), anti-acne drugs, topical and oral retinoids, topical antibacterial agents to the face, and any immunosuppressive drugs. Ongoing oral medications not expected to interfere with study assessments are allowed if the subject is on a stable regimen.
14. Subjects who are currently enrolled in another clinical investigation or have been enrolled in an acne trial within a period of 30 days prior to enrollment in this study.
15. Subjects who are pregnant or nursing.
16. Subjects who require electrolysis, waxing, or depilatories on the face during conduct of the study.
17. Subjects viewed by the investigator as not being able to complete the study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2007-10; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Paller, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Department of Dermatology, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants in this study were patients clinically diagnosed with acne vulgaris. Participants will be recruited from the clinic. Patients were 18 to 35 years of age with mild to moderate acne vulgaris symmetrical in appearance on both sides of the face.
Groups:
- Subjects: Each subject was randomized to applied benzoyl peroxide 2.5% cream formulation to one side of the face and benzoyl peroxide 2.5% cream formulation plus moisturizer to the other side of the face.
Period: Overall Study
Arm/Group | Subjects
Started | 11
Completed | 10
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Subjects
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Subject Reported Change From Baseline Scale
Description: -1=worse 0=unchanged
  * 1=mild improvement
  * 2=moderate improvement
  * 3=clear
Time Frame: baseline and 1 month
Measure: Number; unit: Participants
Arm/Group | Benzoyl Peroxide 2.5% Cream | Benzoyl Peroxide 2.5% Cream Plus Moisturizing Lotion
Number analyzed (Participants) | 10 | 10
Participants
  -1=Worse | 0 | 0
  0=Unchanged | 7 | 6
  1=Mild Improvement | 1 | 1
  2=Moderate Improvement | 1 | 2
  3=Clear | 1 | 1

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Benzoyl Peroxide 2.5% | Benzoyl Peroxide 2.5% Plus Moisturizing Lotion
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 11/11 | 6/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benzoyl Peroxide 2.5% (N=11) | Benzoyl Peroxide 2.5% Plus Moisturizing Lotion (N=11)
Dryness (Skin and subcutaneous tissue disorders) | 6 (10) | 2 (3)
Burning (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3)
Itching (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No